CLINICAL TRIAL: NCT05333926
Title: A Prospective, Open-Label Study of Mahana™ IBS, a Smartphone-Delivered Cognitive Behavioral Therapy (CBT) Treatment, in Young Adults Aged 18-21 Years Old With Irritable Bowel Syndrome
Brief Title: MHNA-001 for Young Adults With IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHNA-001-003
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MHNA-001 (Experimental)
  Interventions: Device: MHNA-001

INTERVENTIONS:
Device: MHNA-001 — 3-month digital therapy program designed to reduce the severity of IBS symptoms
  Other Names: Mahana™ for IBS

SUMMARY:
The main objective of this prospective, open-label, non-significant risk study is to assess the efficacy and safety of Mahana™ IBS together with care as usual in approximately 100 young adults with Irritable Bowel Syndrome.

DETAILED DESCRIPTION:
Following informed consent, all participants will complete a series of screening questionnaires to determine eligibility for study entry. Eligible participants will be enrolled, and will receive access to MHNA-001 (Mahana™ for IBS). Participants will use MHNA-001 for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant meets IBS diagnostic criteria via Rome IV questionnaire.
* Participant has IBS, based on IBS-SSS score of ≥125 at time of screening (corresponding to mild, moderate, or severe IBS).
* Participant is 18-21 years of age at the time of consent.
* Participant is able to speak, read, and understand English.
* Participant is capable and willing to complete questionnaires, track symptoms, and complete exercises associated with use of Mahana™ IBS.
* Participant has unrestricted access to an iOS (running iOS 13 or later) or Android smartphone with internet connectivity and sufficient space for Mahana™ IBS to be installed.
* If participant is taking any prescription IBS-related concomitant medications, he/she must have been on a stable dose/regimen for at least 30 days prior to the date of Screening/Enrollment and is not intended to make changes to dose or regimen during the treatment period (i.e., through Week 12 of the study).

Exclusion Criteria:

* Participant has a medical or psychiatric comorbidity that might account for GI symptoms, confound the measurement of IBS symptoms, or compromise the participant's ability to complete the study (ex. inflammatory bowel disease, chronic liver disease, substance abuse disorder, etc.) in the opinion of the investigator.
* Participant is currently using opioids or plans to use for chronic pain management and/or recreation.
* Participant has been hospitalized for psychiatric reasons within 12 months prior to screening.
* Participant is currently experiencing high depression symptom severity as indicated by a score >14 on the PHQ-8.
* Participant is currently experiencing suicidal ideation as indicated by a score of 2 or 3 on item 9 of the Beck Depression Index (BDI). *
* Participant is currently using any prescription digital therapeutic that delivers components of cognitive-behavioral therapies.
* Participant has undergone CBT, any other skills-based, or GI-specific psychological therapy (e.g. Dialectical Behavioral Therapy, Acceptance and Commitment Therapy, Behavioral Activation, Problem-solving Therapy, Gut-Directed Hypnotherapy, etc.) within 2 years of study entry.
* Participant has participated in any investigational trial within 30 days prior to Screening or plans to participate in another clinical trial during the study period.
* Participant is currently pregnant or nursing.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 194 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Change in IBS Severity Scoring System from Baseline to Week 12 | 12 Weeks
  The IBS Severity Scoring System (IBS-SSS) is a validated, 5-item tool for measuring the severity of IBS symptoms in adults with IBS. The survey asks respondents to rate the severity and frequency of their abdominal pain, severity of abdominal distension, stool frequency and consistency, satisfaction with their bowel habits, and interference of IBS with life in general in the last 10 days using a 100-point visual analogue scale. Scores range from 0 to 500 with higher scores indicating more severe IBS symptoms. Mean score changes of 50 points or more over a 3-month period are predictive of a clinically significant improvement

SECONDARY OUTCOMES:
Subject's Global Assessment of Relief at Week 12 | 12 Weeks
  The SGA will be completed by participants at the end of treatment (Week 12). Participants rate their relief from IBS symptoms on a scale of 1 (completely relieved) to 5 (worse). Participants scoring from 1 to 3 are considered responders and those scoring 4-5 are considered non-responders.

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Institute for Clinical Research, Fayetteville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided